CLINICAL TRIAL: NCT03964610
Title: Multimodal Retinal Imaging of Cerebrovascular Stroke
Acronym: OCTAV
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: RHE_2019_10
Record Dates: First submitted 2019-05-24; First posted 2019-05-28 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Stroke; Cerebrovascular Accidents
Keywords: optical coherence tomography (OCT-A); color fundus photography (CFP); Retinal microvascularization; Cerebral microangiopathy
MeSH Terms: conditions — Stroke; Cerebral Small Vessel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: color fundus photography (CFP) and OCT-A — Included patients will have an ophthalmologic assessment (OCT-A and CPF) after stabilization and at 3 months follow-up.

SUMMARY:
The hypothesis is that in patients with stroke, abnormalities of retinal microvascularization shown on color fundus photography and the depletion of retinal capillary density evaluated by OCT-A are markers of acute impairment of microcirculation of the central nervous system and are correlated with lesions on brain imaging.

Patients hospitalized for stroke MRI-confirmed, will be included. An ophthalmologic assessment including color fundus photography (CFP) and OCT-A will be carried out after stabilization and at 3 months follow-up. Outcomes assessor will be blinded.

ELIGIBILITY:
Inclusion criteria:

* Acute ischemic stroke
* With cerebral microangiopathy (defined by a SVD score > 1)

Exclusion criteria:

* Acute hemorrhagic stroke
* Anophthalmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute patients with a stroke will be included
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Presence of an anomaly in color fundus photography or an anomaly of retinal capillary density to OCT-A | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation A de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No